CLINICAL TRIAL: NCT04704544
Title: Effectiveness of Tele-rheumatology for Delivering High Quality Rheumatology Care During the COVID-19 Crisis
Brief Title: Effectiveness of Tele-rheumatology for Delivering High Quality Rheumatology Care During the COVID-19 Crisis (EVOLVE)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of California, San Francisco (Other); Tulane University (Other); Rheumatology Research Foundation (Other)
Responsible Party: Principal Investigator, Maria Danila, MD, MSc, MSPH, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300006553; 0000000 (Other: Rheumatology Research Foundation)
Record Dates: First submitted 2021-01-06; First posted 2021-01-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Rheumatic Diseases
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: We will conduct an open label, two-period, multi-center, non-inferiority, patient-level randomized controlled trial comparing tele-rheumatology (audio +/- video) with usual care (in-person) visits. Patients will be randomized to the sequence of care for their next two visits (V1 and V2): i) tele-rheumatology (V1) + usual care (V2), OR ii) usual care (V1) + tele-rheumatology (V2). Primary outcome will be ascertained after the first visit (V1).
Who Masked: Care Provider
Masking Description: Providers will be masked to the random assignment of participant visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tele-rheumatology first visit and Usual Care second visit (Experimental): Participants randomized to this visit will receive a tele-rheumatology visit first.
  Interventions: Other: Tele-rheumatology
- Usual Care first visit and Tele-rheumatology second visit (Experimental): Participants randomized to this visit will receive a usual care visit first.
  Interventions: Other: Tele-rheumatology

INTERVENTIONS:
Other: Tele-rheumatology — Participants will receive virtual visits via video conferencing and/or phone.

SUMMARY:
While tele-rheumatology (TR) visits are a COVID-19 related necessity, there is a lack of rigorous data on the comparative effectiveness of TR versus (vs) in-person usual care (UC) especially in medically at-risk populations such as people with rheumatic and musculoskeletal disease (RMD) using immunosuppressive drugs (IS). This clear research gap was highlighted by the American College of Rheumatology in its recent Task Force Report on Telehealth in the COVID era. In this study, the investigators will rigorously evaluate the comparative effectiveness of TR visits for high risk people living with RMD and among those from socially vulnerable populations, in the COVID-19 era. This study is of key public health importance and relevance to rheumatology since it addresses the urgent clinical and policy needs to provide safe, efficacious, and equitable care to diverse patients with RMD during and beyond the COVID-19 crisis. Our proposal is very responsive to the RRF's Notice of Special interest on COVID-19 in improving the care of people with RMD during the COVID-19 pandemic. The investigators will perform the first randomized experiment of tele-rheumatology, generating high quality evidence to guide the use of this technology across diverse populations of people with RMDs. Beyond the high public health impact of this study for people with RMDs, the investigators expect that our findings will have high generalizability to other at-risk patient populations with multimorbidity and inform rheumatology practice into the foreseeable future.

DETAILED DESCRIPTION:
People with RMDs, especially those with multi-comorbidities and on IS are among the most at-risk for COVID-19-related fragmented care and poor outcomes. RMD burden is high in terms of disability-adjusted-life years (DALYs) and has been escalating. Beyond the prevailing challenges to in-person visits such as scheduling conflicts, transportation, or disability, the COVID-19 pandemic has further exacerbated RMD patient burden through disruptions in healthcare delivery (e.g. limited availability of in-person visits). Thus, high quality adaptations of healthcare services for people living with RMD including through TR in the context of the COVID-19 crisis are badly needed. The investigators found from a recent survey of 24,500 people living with RMD that 60% of respondents avoided in-person clinic visits. However, with the increasing availability of technology (90% Americans have internet access, 81% are online daily most patients and clinicians can engage in some form of TR. Due to widespread social distancing and major health policy changes necessitated by COVID-19, TR has been swiftly adopted (but minimally tested) as a means to deliver ongoing care for people with RMD. Because patients can be evaluated in their own homes, thus avoiding travel that increases COVID-19 risk, this approach provides means of healthcare for socially and medically vulnerable groups, such as those residing in rural areas and those with comorbidities, a group particularly at high risk of COVID-19 complications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatic disease (e.g. rheumatoid arthritis, SLE)

Exclusion Criteria:

* unstable rheumatic disease that needs in-person visits (e.g. recent diagnosis of severe lupus nephritis)
* expected in-office procedures (e.g., joint injection)
* lack of access to phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 36-72 hours post visit after the first visit
  Patient satisfaction with type visit. Assessed with AHRQ's Consumer Assessment of Healthcare Providers and Systems (CAHPS)® survey

SECONDARY OUTCOMES:
Patient preference | 36-72 hours post visit, after the second visit
  Patient preference with type visit. Assessed using "If you had a choice, what type of visit would you prefer?" with options a. telemedicine, b. in-office

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman CH, Ramsey-Goldman R. Widening Disparities Among Patients With Rheumatic Diseases in the COVID-19 Era: An Urgent Call to Action. Arthritis Rheumatol. 2020 Sep;72(9):1409-1411. doi: 10.1002/art.41306. Epub 2020 Aug 9. No abstract available. PMID 32379381
- [Background] Brooks PM. The burden of musculoskeletal disease--a global perspective. Clin Rheumatol. 2006 Nov;25(6):778-81. doi: 10.1007/s10067-006-0240-3. Epub 2006 Apr 12. PMID 16609823
- [Background] Donelan K, Barreto EA, Sossong S, Michael C, Estrada JJ, Cohen AB, Wozniak J, Schwamm LH. Patient and clinician experiences with telehealth for patient follow-up care. Am J Manag Care. 2019 Jan;25(1):40-44. PMID 30667610
- [Background] Michaud K, Wipfler K, Shaw Y, Simon TA, Cornish A, England BR, Ogdie A, Katz P. Experiences of Patients With Rheumatic Diseases in the United States During Early Days of the COVID-19 Pandemic. ACR Open Rheumatol. 2020 Jun;2(6):335-343. doi: 10.1002/acr2.11148. Epub 2020 May 9. PMID 32311836
- [Background] Webster P. Virtual health care in the era of COVID-19. Lancet. 2020 Apr 11;395(10231):1180-1181. doi: 10.1016/S0140-6736(20)30818-7. No abstract available. PMID 32278374
- [Background] Bachireddy C, Chen C, Dar M. Securing the Safety Net and Protecting Public Health During a Pandemic: Medicaid's Response to COVID-19. JAMA. 2020 May 26;323(20):2009-2010. doi: 10.1001/jama.2020.4272. No abstract available. PMID 32191260
- [Background] Uscher-Pines L, Fischer S, Tong I, Mehrotra A, Malsberger R, Ray K. Virtual First Responders: the Role of Direct-to-Consumer Telemedicine in Caring for People Impacted by Natural Disasters. J Gen Intern Med. 2018 Aug;33(8):1242-1244. doi: 10.1007/s11606-018-4440-8. No abstract available. PMID 29691713
- [Background] Hayes BL, Curtis JR, Laster A, Saag K, Tanner SB, Liu C, Womack C, Johnson KC, Khaliq F, Carbone LD. Osteoporosis care in the United States after declines in reimbursements for DXA. J Clin Densitom. 2010 Oct-Dec;13(4):352-60. doi: 10.1016/j.jocd.2010.08.001. PMID 21029972
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Nesbitt TS, Marcin JP, Daschbach MM, Cole SL. Perceptions of local health care quality in 7 rural communities with telemedicine. J Rural Health. 2005 Winter;21(1):79-85. doi: 10.1111/j.1748-0361.2005.tb00066.x. PMID 15667014
- [Background] Yang J, Zheng Y, Gou X, Pu K, Chen Z, Guo Q, Ji R, Wang H, Wang Y, Zhou Y. Prevalence of comorbidities and its effects in patients infected with SARS-CoV-2: a systematic review and meta-analysis. Int J Infect Dis. 2020 May;94:91-95. doi: 10.1016/j.ijid.2020.03.017. Epub 2020 Mar 12. PMID 32173574
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076